CLINICAL TRIAL: NCT04389918
Title: A Phase I Study of the Tolerability/Palatability of TalityTM Synthetic Meal Replacement in Patients With Prostate Cancer
Brief Title: Tolerability/Palatability of TalityTM Synthetic Meal Replacement in Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Filtricine Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-55337; PROS0100 (Other: OnCore); IRB-55337 (Other: Stanford IRB)
Record Dates: First submitted 2020-05-11; First posted 2020-05-15 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tality (Experimental): Participants will receive TalityTM as their sole intake for nutritional purposes for a 4 week period.
  Interventions: Other: Tality

INTERVENTIONS:
Other: Tality — Synthetic meal replacements, delivered in many varieties of 400 kCal packets, Manufacturer: Filtricine, Inc.

SUMMARY:
This study will find out if a meal replacement of this type is satisfying and tolerable for men with prostate cancer. Participants will receive meal replacements of TalityTM as their expected sole source of nutrition for 4 weeks. The purpose of the study is to test whether TalityTM Synthetic Meal Replacements are suitable to be used in larger studies of patients with prostate or other types of cancer.

DETAILED DESCRIPTION:
Primary Objective: Determine the appeal/tolerability/palatability of a diet consisting solely of TalityTM synthetic meal replacement in participants with prostate cancer Secondary Objective: Evaluate the effect of TalityTM on safety parameters including laboratory tests, nutritional status and adverse effects

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven prostate cancer with stable or rising PSA levels, defined as three consecutive PSA levels, each value greater than 1 week apart, with fluctuation between the three values no more than 10% downward. The third PSA needs to be within 30 days prior to enrollment and >= 0.1.
* Patients may previously have been on any regimen of chemotherapy completed at least one month prior. Patients may be on any stable form of anti-androgen therapy.
* Males >= age 18.
* All patients must have a life expectancy of > 6 months.
* Patients must have an ECOG Performance Status of <= 1
* Patients must have no clinically significant abnormalities of organ or bone marrow function
* Patients must have the ability to understand and the willingness to sign a written informed consent document, and the willingness/ability to comply with the protocol activities.

Exclusion Criteria:

* Chemotherapy within one month prior to enrollment or plans to receive chemotherapy within one month after enrollment. Patients who are expected to require new or modified anti-androgen therapy during the course of the study are also excluded.
* Patients may not be receiving any other Investigational Agents during the course of the study.
* Patients who experience frequent symptoms of a gastrointestinal nature (e.g., diarrhea, abdominal bloating, constipation or pain) are excluded.
* Known CNS metastases.
* Patients who, in the opinion of the Principal Investigator, have a clinically significant co-morbid disease that is likely to affect the ability of the patient to complete the trial, interfere with their ability with measurement of self-reported outcomes or result in adverse events unrelated to TalityTM are excluded.
* Patients with a history of food allergy are excluded.
* Concomitant medications necessary to treat baseline disorders are allowed (e.g., hypertension, diabetes, and hyperlipidemia).
* Patients requiring concomitant medications that, in the opinion of the Principal Investigator, have an unacceptable risk of adverse effects due to their nature (e.g., anti-coagulant therapy, immuno-modulatory agents for autoimmune disease) must be excluded.
* Pregnant or nursing patients will not be enrolled since prostate cancer is limited to males.
* HIV-positive patients with active infections, HIV related cancer or poorly controlled viral loads must be excluded. HIV-positive patients who are stable on anti-viral therapy may be enrolled.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Proportion of Completers | 4 weeks
  The proportion of participants who complete the 4 week study using TalityTM as their sole source of nutrition at a high level of adherence (75% of days, 21+ days out of the 28 day study).

SECONDARY OUTCOMES:
Change in weight from baseline | 4 weeks
  Change in weight will be measured from baseline.
Change in amino acid levels | 4 weeks
  Change in amino acid levels as compared to baseline will be measured. The following amino acids will be analyzed a-Aminoadipic Acid, a-Aminobutyric Acid, Alanine, Arginine, Asparagine, Aspartic Acid, b-Alanine, b-Aminoisobutyric Acid, Citrulline, Cystathionine, Cystine, Ethanolamine, Glutamic Acid, Glutamine, Glycine, Histidine, Homocystine, Hydroxyproline, Isoleucine, Leucine, Lysine, Methionine, Ornithine, Phenylalanine, Proline, Sarcosine, Serine, Taurine, Threonine, Tryptophan, Tyrosine, Valine. It will be measured in micro-moles per Liter.
Change in Prostate Specific Antigen | 4 weeks
  Change from baseline in the serum level of prostate specific antigen (PSA).

CONTACTS AND LOCATIONS:
Overall Officials: Randall S Stafford, MD, PhD, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No